CLINICAL TRIAL: NCT05635110
Title: A Phase 1, Open-label Drug-drug Interaction Study to Evaluate the Effects of Omeprazole and Rifampin on the Pharmacokinetics of VX-548 in Healthy Subjects
Brief Title: Evaluation of the Effects of Omeprazole and Rifampin on the Pharmacokinetics of VX-548 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: VX22-548-013
Record Dates: First submitted 2022-11-22; First posted 2022-12-02 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Omeprazole; Rifampin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A (Experimental): Participants will receive a single dose of VX-548 on Day 1 and a single dose of omeprazole once daily (qd) on Days 10 through Day 12. On Day 13, participants will receive omeprazole followed by VX-548 under fasted conditions.
  Interventions: Drug: VX-548; Drug: Omeprazole
- Part B (Experimental): Participants will receive a single dose of VX-548 on Day 1 followed by rifampin qd on Days 10 through Day 27. On Day 19, participants will be co-administered rifampin and VX-548 under fasted conditions.
  Interventions: Drug: VX-548; Drug: Rifampin

INTERVENTIONS:
Drug: VX-548 — Tablets for oral administration.
  Other Names: Suzetrigine
Drug: Omeprazole — Tablets for oral administration.
  Arms: Part A
Drug: Rifampin — Capsules for oral administration.
  Arms: Part B

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics and safety of VX-548 and its metabolite in the absence and presence of omeprazole or rifampin, in healthy participants.

DETAILED DESCRIPTION:
This clinical trial information was submitted voluntarily under the applicable law and, therefore, certain submission deadlines may not apply. (That is, clinical trial information for this applicable clinical trial was submitted under section 402(j)(4) (A) of the Public Health Service Act and 42 CFR 11.60 and is not subject to the deadlines established by sections 402(j)(2) and (3) of the Public Health Service Act or 42 CFR 11.24 and 11.44.).

ELIGIBILITY:
Key Inclusion Criteria:

* Body mass index (BMI) of 18.0 to 32.0 kilogram per meter square (kg/m^2)
* A total body weight greater than (>) 50 kg

Key Exclusion Criteria:

* History of febrile illness or other acute illness that has not fully resolved within 14 days before the first dose of study drug
* Any condition possibly affecting drug absorption
* History of cardiovascular disease
* Participants of child-bearing potential

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2023-06-08 (Actual); Study Completion 2023-06-08 (Actual)

PRIMARY OUTCOMES:
Part A: Maximum Observed Plasma Concentration (Cmax) of VX-548 and its Metabolite in the Absence and Presence of Omeprazole | Day 1 up to Day 22
Part A: Area Under the Concentration Versus Time Curve From the Time of Dosing Extrapolated to Infinity (AUC0-inf) of VX-548 and its Metabolite in the Absence and Presence of Omeprazole | Day 1 up to Day 22
Part B: Maximum Observed Plasma Concentration (Cmax) of VX-548 and its Metabolite in the Absence and Presence of Rifampin | Day 1 up to Day 28
Part B: Area Under the Concentration Versus Time Curve From the Time of Dosing Extrapolated to Infinity (AUC0-inf) of VX-548 and its Metabolite in the Absence and Presence of Rifampin | Day 1 up to Day 28

SECONDARY OUTCOMES:
Part A:Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Day 1 through Safety Follow-up Visit (up to 28 days)
Part B: Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Day 1 through Safety Follow-up Visit (up to 34 days)

CONTACTS AND LOCATIONS:
Locations (1):
- CMAX Clinical Research, Adelaide, Australia

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent-research/clinical-trial-data-sharing